CLINICAL TRIAL: NCT01579643
Title: Randomized Clinical Trial of OCT-guided Laser-assisted Lamellar Anterior Keratoplasty in Children
Brief Title: OCT-guided LALAK in Children
Acronym: LALAK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, Bibiana Jin Reiser, MD: Assistant Professor of Clinical Ophthalmology, Children's Hospital Los Angeles
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB#00006612 LALAK Child
Record Dates: First submitted 2012-01-03; First posted 2012-04-18 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Corneal Opacity
Keywords: cornea; opacity; congenital
MeSH Terms: conditions — Corneal Opacity; Corneal Diseases | interventions — Keratoplasty, Penetrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LALAK (Experimental)
  Interventions: Procedure: OCT guided laser-assisted lamellar anterior keratoplasty (LALAK)
- Penetrating Keratoplasty (KP) (Active Comparator)
  Interventions: Procedure: Penetrating Keratoplasty (KP)

INTERVENTIONS:
Procedure: OCT guided laser-assisted lamellar anterior keratoplasty (LALAK) — 1. The top hat-shaped donor cornea graft with tapered brim will be cut using a femtosecond (fs) laser at the eye bank. An anterior diameter of 6.0 mm will be used. The depth of the anterior side cut will match the planned excimer ablation depth.
  2. The host cornea bed will be prepared with an excimer laser.
  3. Descemet's membrane will be peeled off the graft, and the graft sutured into the host bed.
  Arms: LALAK
Procedure: Penetrating Keratoplasty (KP) — 1. A trephine is used to perform a full thickness cut of a round area of cornea from the both patient's and donor's cornea.
  2. The donor cornea is then sutured where the patient's cornea was.
  Arms: Penetrating Keratoplasty (KP)

SUMMARY:
The primary goal of the trial is to determine if laser-assisted lamellar anterior keratoplasty (LALAK) will reduce the risks of post-operative complications such as adhesions, glaucoma and cataract that are associated with pediatric penetrating keratoplasty (PK).

DETAILED DESCRIPTION:
There is a great need for lamellar keratectomy in the treatment of congenital opacities because the rejection rate in pediatric PK is 4-5 times higher than in adults. In addition, the intraocular inflammatory reaction in infants often leads to synechiae, glaucoma, and cataract. Because LALAK does not penetrate the eye and preserves the host endothelium, it could reduce the risk of these complications. Keratoplasty must be performed at this early age to prevent amblyopia.

In this study, OCT-guided LALAK will be performed in patients whose vision is limited by opacity in the anterior 2/3 of the cornea. The objective is to determine if LALAK will provide an equal or better visual outcome than traditional PK without the associated post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Vision limited by opacity in the anterior 2/3 of the corneal stroma
* Posterior opacity and endothelial defect must be less than 1 mm in diameter

Exclusion Criteria:

* Presence of cataract
* Presence of adhesions of the iris or lens to the cornea
* Inability/unwillingness of parents to give informed consent
* Inability of parents to commit to required visits to complete the study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2012-01; Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Number of LALAK patients with post operative complications compared to PK patients | 24 months
  Results of PK and LALAK will be compared in terms of corneal clarity, graft rejection, intraocular pressure, and vision (if measurable).

CONTACTS AND LOCATIONS:
Overall Officials: Bibiana Reiser, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital of Los Angeles, Los Angeles, California, United States